CLINICAL TRIAL: NCT05364385
Title: Intra-tracheal Instillation of Budesonide Along With Surfactant in Preterm Infants to Prevent Chronic Lung Disease
Brief Title: Intra-tracheal Instillation of Budesonide to Prevent Chronic Lung Disease
Acronym: STOPCLD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1811108822
Record Dates: First submitted 2022-05-02; First posted 2022-05-06 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Infant, Extremely Premature; Acute Lung Injury; Chronic Lung Disease of Prematurity; Budesonide
MeSH Terms: conditions — Acute Lung Injury; Bronchopulmonary Dysplasia | interventions — Budesonide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- S/B group- infants (Experimental): Infants randomized to the study group (S/B group) will receive surfactant and Budesonide - 0.5 mg -1mL
  Interventions: Drug: Infants in the study group (S/B group) will receive surfactant 2.5 mls/kg and Budesonide 0.5 mg (1mL)
- S/P group- control / placebo comparator (Placebo Comparator): Infants randomized to the control group (S/P group) will receive surfactant and placebo (Normal Saline -1mL)
  Interventions: Drug: Infants in the control group (S/P group) receive placebo (Normal saline 1mL)

INTERVENTIONS:
Drug: Infants in the study group (S/B group) will receive surfactant 2.5 mls/kg and Budesonide 0.5 mg (1mL) — Infants in the study group (S/B group) will receive surfactant 2.5 mls/kg and Budesonide 0.5 mg (1mL)
  Other Names: Pulmicort
  Arms: S/B group- infants
Drug: Infants in the control group (S/P group) receive placebo (Normal saline 1mL) — Infants in the control group (S/P group) will receive surfactant 2.5 mls/kg and placebo (Normal saline 1mL)
  Arms: S/P group- control / placebo comparator

SUMMARY:
Preterm infants are randomized to received either Intra-tracheal instillation of budesonide using surfactant as vehicle or a placebo. Intra-tracheal instillation of budesonide using surfactant as vehicle would facilitate its delivery to the periphery of the lung and would inhibit lung inflammation and mitigate acute lung injury.

DETAILED DESCRIPTION:
In extremely premature infants who are ventilated there is ongoing lung injury & lung inflammation. This can perpetuate the need for ongoing ventilation and these infants spend much longer in the hospital. The likelihood of chronic lung disease in this susceptible group is very high and they would need oxygen at home. Surfactant instillation has reduced the need for prolonged mechanical ventilation and to an extent the incidence of chronic lung disease (CLD). But many infants develop CLD and need prolonged oxygen treatment, diuretics and inhaled steroids to suppress the inflammation and obstruction of the airways. Some of the severely affected infants need orally administered steroids. The Inestigators propose to provide a dose of steroids instilled along with the surfactant in the very first day of life so as to prevent the vicious and ongoing cascade of lung injury and inflammation. As it is a poorly absorbed steroid and as only one or two doses is proposed to be used there is no effects within the body and it works locally within the lung. This is hoped to reduce CLD and improve long term outcomes. The population most susceptible to CLD is the extreme preterm infant with RDS who needs mechanical ventilation soon after birth. One of the groups will receive the surfactant with saline and the other group will receive the surfactant along with topical steroid. The groups will be followed during the hospital stay. survival along with duration of ventilation, duration of hospital stay and oxygen needs are noted. To study the hoped for long term benefits the investigators would note the long term neuro-development - if they were followed as per hospital policy between 18 months and 26 months. Intra-tracheal instillation of budesonide using surfactant as vehicle would facilitate its delivery to the periphery of the lung and would inhibit lung inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at < 30+0/7 weeks (23+0 - 29+6/7) gestational age (GA) OR with preterm infants with a birth weight (BW) which is < 1500 gm AND if they have severe respiratory distress syndrome (RDS) (Clinical diagnosis based on the need for mechanical ventilation in preterm infant or if they have radiologic features of RDS along with need for positive distending airway pressure and fractional inspired oxygen (FiO2) > 0.3)

Exclusion Criteria:

1. major congenital defects
2. chromosomal abnormality
3. pneumothorax
4. Known surgical disease
5. Known or suspected congenital heart disease
6. Infant not considered viable by physician
7. Severe sepsis / infections
8. Likely to be extubated within the next 24 hours

Max Age: 18 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change of combined inflammatory cytokines | 4 weeks
  Change in inflammatory cytokines /chemokines (interleukin-6, 8, 10 and Tumor Necrosis Factor α (TNF-α) levels

SECONDARY OUTCOMES:
chronic lung disease | 36 weeks corrected gestational age (CGA)
  Supplemental oxygen requirement at 36 weeks corrected gestational age
Mortality | upto 40 weeks corrected gestational age (CGA)
  All cause mortality
Ventilator days | Upto 40 weeks corrected gestational age (CGA)
  duration of ventilation
Neuro-developmental outcome | 18 - 26 months corrected postnatal age
  Composite Bailey III neuro-developmental score. Scores range overall from 40 to 160 and for Cognitive: 55-145; Language: 47-153; Motor: 46-154; Social-Emotional: 55-145 with lower score for poor outcome and higher score for better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided